CLINICAL TRIAL: NCT00519896
Title: Phase II Study of Sunitinib in Iodine Refractory Differentiated Thyroid Cancer and Metastatic Medullary Carcinoma of Thyroid With Functional Imaging Correlation
Brief Title: Sunitinib Malate in Treating Patients With Iodine-Refractory Recurrent or Metastatic Thyroid Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Renato Martins, Principal Investigator, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6494; NCI-2011-01305 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2007-08-21; First posted 2007-08-23 (Estimated); Results first posted 2017-04-25 (Actual); Last update posted 2017-04-25 (Actual); Status verified 2017-01

CONDITIONS: Recurrent Thyroid Cancer; Stage IVA Follicular Thyroid Cancer; Stage IVA Papillary Thyroid Cancer; Stage IVB Follicular Thyroid Cancer; Stage IVB Papillary Thyroid Cancer; Stage IVC Follicular Thyroid Cancer; Stage IVC Papillary Thyroid Cancer; Thyroid Gland Medullary Carcinoma
MeSH Terms: conditions — Thyroid Neoplasms; Adenocarcinoma, Follicular; Thyroid Cancer, Papillary; Carcinoma, Medullary | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (enzyme inhibitor therapy, antiangiogenesis therapy) (Experimental): Patients receive sunitinib malate PO QD. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: sunitinib malate

INTERVENTIONS:
Drug: sunitinib malate — Given PO
  Other Names: SU11248; sunitinib; Sutent

SUMMARY:
This phase II trial studies how well giving sunitinib malate works in treating patients with iodine-refractory recurrent or metastatic thyroid cancer. Sunitinib malate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth or by blocking blood flow to the tumor

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the response of sunitinib (sunitinib malate) per Response Evaluation Criteria in Solid Tumors (RECIST) criteria in patients with recurrent/metastatic iodine refractory well differentiated thyroid carcinoma (WDTC) or medullary thyroid carcinoma (MTC).

SECONDARY OBJECTIVES:

I. Evaluate early positron emission tomography (PET) changes in patients with WDTC and MTC treated with sunitinib.

II. Determine the safety and toxicity of sunitinib given as a continuous treatment in patients with WDTC and MTC.

III. Evaluate the effect of sunitinib therapy on overall survival, duration of response and time-to-progression.

IV. Evaluate serial tumor markers, thyroglobulin (WDTC) or calcitonin (MTC), during therapy. These measurements will not be used to define disease progression or response.

V. Correlate changes in serial tumor markers with radiologic response.

OUTLINE:

Patients receive sunitinib malate orally (PO) once daily (QD). Treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven metastatic WDTC or MTC
* Evidence of refractoriness to iodine therapy for WDTC documented by a combination of imaging and thyroglobulin or by biopsy
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 3
* Evidence of fludeoxyglucose F 18 (FDG) PET avid metastatic tumors
* Measurable disease by RECIST criteria
* Resolution of all acute toxic effects of prior systemic therapy (including iodine therapy or chemotherapy), radiotherapy or surgical procedure to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0 grade =< 1
* Total serum bilirubin =< 1.5 x upper limit of normal (ULN) (patients with Gilbert's disease exempt)
* Serum transaminases =< 2.5 x ULN or =< 5.0 X ULN if secondary to liver metastases
* Serum creatinine =< 1.5 x ULN
* Absolute neutrophil count (ANC) >= 1.5 X 10^9/L
* Platelets >= 100,000/uL
* Hemoglobin >= 9.0 g/dL
* Willingness and ability to comply with scheduled visits, treatment plans and laboratory tests and other study procedures
* Male and female patients with reproductive potential must use an acceptable contraceptive method
* Signed and dated informed consent document indicating that the patient has been informed of all the pertinent aspects of the trial prior to enrollment

Exclusion Criteria:

* Concomitant treatment in another therapeutic clinical trial
* ECOG performance status >= 3
* Symptomatic, untreated, brain metastasis
* Second primary malignancy that is clinically detectable or clinically significant at the time of consideration for study enrollment
* Full-dose anticoagulation defined as:

  * Low molecular weight heparin use with the intent of full dose anticoagulation; example: enoxaparin 1.5 mg/kg daily or equivalent
  * Warfarin use to keep international normalized ratio (INR) greater than or equal to 2
* History of gross hemoptysis (defined as bright red blood of at least 1/2 teaspoon or 2.5 mL per episode) within 3 months prior to study drug administration unless definitively treated with surgery or radiation
* Any of the following within the 6 months prior to study drug administration: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack, or pulmonary embolism; ongoing cardiac dysrhythmias of NCI CTCAE Version 3.0 grade >= 2
* Type I Diabetes Mellitus; patients with Type II Diabetes Mellitus will be included as long as their glucose can be controlled between levels of 80 and 150 mg/dL
* Uncontrolled Hypertension (> 150/100 mm Hg despite optimal medical therapy)
* Major surgery or radiation therapy within 4 weeks of starting the study treatment
* Other severe acute or chronic medical or psychiatric condition, or laboratory abnormality that would impart, in the judgment of the investigator, excess risk associated with study participation or study drug administration, or which, in the judgment of the investigator, would make the patient inappropriate for entry into this study
* Pregnancy or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2007-07; Primary Completion 2015-05 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Renato Martins, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Enzyme Inhibitor Therapy, Antiangiogenesis Therapy)
Started | 35
Completed | 33
Not Completed | 2
Not completed — Protocol Violation | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: All 35 patients that signed consent and received at least one dose of study therapy are included.
Arm/Group | Treatment (Enzyme Inhibitor Therapy, Antiangiogenesis Therapy)
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 8
Age, Continuous [Median (Full Range); unit: years] | 61 [34 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 17
Region of Enrollment [Number; unit: participants]
  United States | 35

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.",
Time Frame: At baseline until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Enzyme Inhibitor Therapy, Antiangiogenesis Therapy)
Number analyzed (Participants) | 33
Participants | 11

2. Secondary Outcome: Safety and Toxicity of Sunitinib Malate Given as a Continuous Treatment Rated for Toxicity Using the NCI Common Toxicity Criteria (CTC) Version 3.0
Description: Only adverse events that were grade 3 and higher using NCI Common Toxicity Criteria (CTC) version 3.0 were recorded.
Time Frame: On day 1, monthly while on study treatment, and after completion of study treatmentthrough study completion, an average of 2 years
Population: All patients that received at least one dose of sunitinib malate were included in the analysis.
Measure: Number; unit: participants
Arm/Group | Treatment (Enzyme Inhibitor Therapy, Antiangiogenesis Therapy)
Number analyzed (Participants) | 35
participants
  Fatigue | 4
  Neutropenia | 12
  Hand/Foot syndrome | 6
  Diarrhea | 6
  Leukopenia | 11
  Gastrointestional Hemorrhage | 1

3. Secondary Outcome: Time-to-tumor Progression Measured From the Date of Enrollment to the First Date of Progression of Disease
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: At 30 days from the last dose of study treatment and then for 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Enzyme Inhibitor Therapy, Antiangiogenesis Therapy)
Number analyzed (Participants) | 33
months | 12.8 [8.9 to NA] — The data collection time period ended before all patients experienced disease progression.

ADVERSE EVENTS:
Time Frame: adverse events were collected from the date of the first dose of sunitinib through 30 days following the last dose of sunitinib or up to 2 years.
Arm/Group | Treatment (Enzyme Inhibitor Therapy, Antiangiogenesis Therapy)
Serious Adverse Events (participants affected / at risk) | 1/35
Other Adverse Events (participants affected / at risk) | 35/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Enzyme Inhibitor Therapy, Antiangiogenesis Therapy) (N=35)
Gastrointestional Bleed (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Enzyme Inhibitor Therapy, Antiangiogenesis Therapy) (N=35)
fatigue (General disorders) | 9 (9)
Dehydration (Gastrointestinal disorders) | 2 (2)
Anorexia (Gastrointestinal disorders) | 1 (1)
Mucositis (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 9 (9)
Nausea/vomiting (Gastrointestinal disorders) | 3 (3)
Odynophagia (Gastrointestinal disorders) | 2 (2)
Gastrointestional Bleed (Gastrointestinal disorders) | 5 (5)
Hand/Foot Syndrome (Skin and subcutaneous tissue disorders) | 9 (9)
Hemoptysis (Blood and lymphatic system disorders) | 2 (2)
Tachycardia (Cardiac disorders) | 2 (2)
Hypertension (Vascular disorders) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 11 (11)
Neutropenia (Blood and lymphatic system disorders) | 12 (12)
anemia (Blood and lymphatic system disorders) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Epistaxis (Blood and lymphatic system disorders) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Neuropathy (Nervous system disorders) | 1 (1)
Infection (Infections and infestations) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes